CLINICAL TRIAL: NCT01313403
Title: Imaging Serotonin 5-HT1A Receptors in the High Affinity State in Brains of Patients With Major Depressive Disorder
Brief Title: Imaging Serotonin 5HT1A Receptors in Patients With Major Depressive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 110097; 11-M-0097
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-25

CONDITIONS: Major Depression; Unipolar Depression; Depression; Anxiety Disorder
Keywords: 5-HT1A Receptors; Major Depression; PET Imaging; Depression; Healthy Volunteer; HV
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Anxiety Disorders | interventions — Antidepressive Agents; Selective Serotonin Reuptake Inhibitors

INTERVENTIONS:
Other: Antidepressant (SSRI)

SUMMARY:
Background:

- Medications to treat major depression act on a brain chemical called serotonin, which binds to receptors on brain cells. More research is needed on how serotonin receptors work in the brain, and imaging studies such as magnetic resonance imaging (MRI) can provide information on how these receptors function in the brains of individuals with depression and healthy volunteers. The experimental radioactive chemical [11C]CUMI has been designed to react with serotonin receptors, and researchers are interested in studying its effectiveness using positron emission tomography (PET) scanning to see how well it gets into the brain.

Objectives:

- To evaluate the effectiveness of the radiotracer [11C]CUMI in brain imaging studies of serotonin receptors.

Eligibility:

- Individuals between 18 and 55 years of age who either have been diagnosed with major depressive disorder or are healthy volunteers.

Design:

* Participants will be screened with a full medical history, physical and psychiatric examination, blood and urine tests, and questionnaires about mood. Participants will also have an electrocardiogram at this visit.
* At the first study visit, participants will have a MRI scan of the brain to provide baseline data on brain function.
* At the second study visit, participants will have a PET scan with the [11C]CUMI contrast agent.
* No treatment will be provided as part of this protocol....

DETAILED DESCRIPTION:
Eighteen million people in the United States are currently suffering from Major Depressive Disorder, which is characterized by episodes of low mood, poor self attitude and poor vitality. Of those suffering from Major Depressive Disorder (MDD), only one third completely improve, but even among these cases, there is a waiting period of several weeks or more during which antidepressants take effect. Our inability to adequately treat MDD is evident in its being ranked number one in Disability Adjusted Life Years (DALY) among persons aged 15-44. Given this profound burden, improving our understanding of the molecular basis of MDD is of utmost importance in the development of novel antidepressant medications.

Serotoninergic neurotransmission is implicated in MDD, as demonstrated by the relative success of selective serotonin reuptake inhibitors (SSRIs). SSRIs block the reuptake of serotonin through the serotonin transporter, which then increases serotonin at the synaptic cleft. Serotonin then binds to 5-HT1A receptors, which are G-protein coupled receptors that are present both presynaptically and postsynaptically. Presynaptically, these receptors act as autoinhibitory receptors, triggering decreased firing rates and serotonin release. This autoinhibition, which lasts for about two weeks, is believed to be the reason why patients experience a delay in symptomatic improvement after initiation of SSRIs. Serotonin binding to postsynaptic receptors mediates symptomatic improvement of depression. Multiple positron emission tomography (PET) studies utilizing antagonists at 5-HT1A have been conducted. The results are mixed, with some noting increased and others noting decreased 5-HT1A in the brains of patients with MDD. While clinical heterogeneity and the effects of previous treatment with SSRIs may be confounding factors, the lack of consistent finding could also be secondary to using antagonist rather than agonist radioligands. Unlike agonists, antagonists are unable to discriminate between 5-HT1A in the high and low affinity states, and only the high affinity state, which is G-protein-coupled, allows for activity at the 5-HT1A receptor.

We propose a PET study using 5-HT1A radiolabelled agonist, C(11)CUMI, to determine whether there is a difference in the density and distribution of 5-HT1A in the high affinity state in the brains of patients with MDD versus controls. We will perform an internal control at 1-5 days after initiation of SSRI to determine whether increased serotonin causes detectable displacement of C(11)CUMI. At 4-8 weeks after initiation of SSRI treatment, we will reimage patients to determine whether there is a change in the density of 5-HT1A in the high affinity state.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with MDD (Inclusion criteria):

1. Subjects must be between 18-55 years old.
2. Subjects must be able and willing to give written informed consent.
3. Subjects must have a DSMIV diagnosis of Major Depressive Disorder (MDD).
4. Subjects must at the time of study enrollment be experiencing an episode of Major Depression per DSMIV criteria, and as demonstrated by a Hamilton Depression Rating Scale (HDRS; 17 item) greater than 18 (Williams, 1988).

Healthy Volunteers (Inclusion criteria):

1. Subjects must be adults between 18-55 years old.
2. Subjects must be able and willing to give written informed consent.
3. Hamilton Depression Rating Scale (HDRS-17 item) less than 8.

EXCLUSION CRITERIA:

Patients with MDD (Exclusion criteria):

1. With the exception of substance abuse and anxiety disorders, any past or current Axis I diagnosis other than Major Depressive Disorder. With regard to substance abuse disorders, we will allow past diagnoses so long as there is no question of substance or alcohol dependence, the patient has not had substance abuse patterns in the year prior to enrollment, and other criteria regarding LSD and ecstasy use are met (see below). We will screen for substance abuse patterns in the year prior to enrollment by excluding heavy alcohol use, as defined as greater than 14 drinks per week for men and greater than 7 drinks per week for women. With regard to anxiety disorders, we will allow past or present diagnoses of Generalized Anxiety Disorder, social phobia and panic disorder, so long as the anxiety disorder is not felt to outweigh the magnitude of the diagnosis of Major Depressive Disorder. This will be determined by clinical investigators in this protocol. Particular attention will be made to ensure that the patient does not have a diagnosis of Bipolar disorder, Schizoaffective disorder or Premenstrual dysphoric disorder (PMDD).
2. Any history of Lysergic acid diethylamide (LSD) use, because it may alter serotonin receptor properties.
3. History of ecstasy use more than 3 times in life, because it may alter serotonin receptor properties.
4. Current suicidality or serious depressive symptoms warranting more intensive management than weekly visits in our psychiatric outpatient clinic
5. Psychiatric symptoms warranting psychotropic medications other than the selected SSRI study drug. The exception to this is infrequent use of benzodiazepine (e.g. lorazepam (Ativan), 0.5-1.0 mg for anxiety). Infrequent is defined here as less often than 3 times per week.
6. In women, irregular menses such that it will not be possible to determine the phase of the cycle. This is because previous data show that the phases of the menstrual cycle may affect 5-HT1A binding by radioligand.
7. Clinically significant laboratory abnormalities.
8. Psychotropic medication use (including benzodiazepines and illicit drugs) during the 21 days (42 days for fluoxetine) prior to the PET scan. The exception would be 1-5 doses of 0.5-1.0mg of benzodiazepine (lorazepam (Ativan)) by mouth, separated by at least 24 hours between doses, for anxiety related to study procedures.
9. Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases, brain masses or lesions > 1cm in diameter.
10. Positive HIV status.
11. Metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
12. Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes.
13. History of fetal alcohol syndrome or other neurodevelopmental disorder.
14. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
15. Positive urine drug screen.
16. Inability to lie flat on camera bed for about 2.5 h
17. History of adverse reaction to the medication that we plan to use in the patient, which will be selected among sertraline (Zoloft), citalopram (Celexa) or escitalopram (Lexapro)
18. Pregnancy at time of scan (BetaHCG will be measured in all female patients within 24 hours of scan and must be negative)

Healthy Volunteers (Exclusion criteria):

1. With the exception of substance abuse, any past or current Axis I diagnosis. With regard to substance abuse disorders, we will allow past diagnoses so long as there is no question of substance or alcohol dependence, the patient has not had substance abuse patterns in the year prior to enrollment, and other criteria regarding LSD and ecstasy use are met (see below).
2. Any history of psychotic symptoms
3. If female, any history of Premenstrual Dysphoric Disorder (PMDD), because PMDD has been shown to correlate with changes in 5-HT1A distribution in brain.
4. Any history of Lysergic acid diethylamide (LSD) use, because it may alter serotonin receptor properties.
5. History of ecstasy use more than 3 times in life, because it may alter serotonin receptor properties.
6. In women, irregular menses such that it will not be possible to determine the phase of the cycle. This is because previous data show that the phases of the menstrual cycle may affect 5-HT1A binding by radioligand.
7. Clinically significant laboratory abnormalities.
8. Psychotropic medication use (including benzodiazepines and illicit drugs) during the 21 days (42 days for fluoxetine/ Prozac, which has a longer half-life) prior to the PET scan.
9. Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases or any cardiopulmonary disease that would increase risks associated with sedation.
10. Positive HIV status.
11. Metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
12. Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes.
13. History of fetal alcohol syndrome or other neurodevelopmental disorder.
14. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
15. Positive urine drug screen.
16. Inability to lie flat on camera bed for about 2.5 h
17. Pregnancy at time of scan (BetaHCG will be measured in all female patients within 24 hours of scan and must be negative)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02-10; Primary Completion 2012-04-25 (Actual); Study Completion 2012-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)

REFERENCES:
- [Background] Alpert JE, Franznick DA, Hollander SB, Fava M. Gepirone extended-release treatment of anxious depression: evidence from a retrospective subgroup analysis in patients with major depressive disorder. J Clin Psychiatry. 2004 Aug;65(8):1069-75. PMID 15323591
- [Background] Amsterdam JD, Brunswick DJ, Gibertini M. Sustained efficacy of gepirone-IR in major depressive disorder: a double-blind placebo substitution trial. J Psychiatr Res. 2004 May-Jun;38(3):259-65. doi: 10.1016/j.jpsychires.2003.10.005. PMID 15003431
- [Background] Amsterdam JD. Gepirone, a selective serotonin (5HT1A) partial agonist in the treatment of major depression. Prog Neuropsychopharmacol Biol Psychiatry. 1992 May;16(3):271-80. doi: 10.1016/0278-5846(92)90079-t. PMID 1350353
- [Background] Artigas F, Romero L, de Montigny C, Blier P. Acceleration of the effect of selected antidepressant drugs in major depression by 5-HT1A antagonists. Trends Neurosci. 1996 Sep;19(9):378-83. doi: 10.1016/S0166-2236(96)10037-0. PMID 8873352